CLINICAL TRIAL: NCT05334303
Title: Prevalence and Prognostic Impact of Epigenetic MMRd in Endometrial Carcinomas
Brief Title: The Impact of Epigenetic MMRd in Endometrial carcinomas-a Real World Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC-KY-KS-2022-105
Record Dates: First submitted 2022-04-07; First posted 2022-04-19 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-03

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- epigenetic MMR deficiency: Tumors with MMR abnormalities by IHC and MLH1 methylation
- probable MMR mutations: Tumors with MMR abnormalities by IHC and without MLH1 methylation
- MMR proficient: without MMR abnormalities by IHC

SUMMARY:
In recent years, the incidence of endometrial carcinoma (EC) has increased significantly and patients tends to be younger. In addition to known risk factors such as obesity, hypertension and diabetes, genetic factors also play an important role in the occurrence and development of EC. Among them, Mismatch Repair Defect (MMR) can produce mutant phenotypes, leading to cancer susceptibility. Although some articles indicated that epigenetic MMRd, one type of MMRd, predicted poor prognosis among endometrial carcinoma patients, hitherto, the clinicopathological significance and prognosis of epigenetic MMRd has not been determined. To date, there are no relevant large-sample data to investigate the prevalence of epigenetic MMRd in Chinese population, as well as the impact on the prognosis of endometrial cancer. In this setting, The purpose of this study was to investigate the prevalence of epigenetic MMRd and its impact on clinicopathology and prognosis on endometrial cancer among Chinese patients.

DETAILED DESCRIPTION:
We conducted a retrospective real-world study of all endometrial carcinoma cases from 2019 to 2022. The inclusion criterion is all patients diagnosed with endometrial cancer in our hospital from 2019 to 2022 and exclusion criteria are those without histological specimens in our hospital. After immunohistochemistry and MLH1-promoter methylation testing, tumors were classified into 3 groups according to status of mismatch repair defects. Tumors with MMR abnormalities by IHC and MLH1 methylation were classified as epigenetic MMR deficiency while those without MLH1 methylation were classified as probable MMR mutations, and those without MMRd were classified as MMR proficient. The first outcome is the prevalence of epigenetic MMRd in endometrial cancer, and the second outcome is Whether the clinicopathological features and prognosis of endometrioid adenocarcinoma differ between the epigenetic MMRd population, MMR proficient population and the Lynch/ Lynch-like population.

ELIGIBILITY:
Inclusion Criteria:

* all patients diagnosed with endometrial cancer in our hospital from 2019 to 2022

Exclusion Criteria:

* those without histological specimens in our hospital

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically confirmed endometrial carcinoma and case slides available for review from 2019 to 2022 in our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-11-17 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of MMRd caused by MLH1 promoter methylation in endometrial carcinoma | up to two years
  the prevalence of epigenetic MMRd in endometrial cancer

SECONDARY OUTCOMES:
progression-free survival time (PFS) | up to two years
  progression-free survival time (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-qiu Lin, Principal Investigator — Department of Gynecologic Oncology, Sun Yat-sen Memorial Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No